CLINICAL TRIAL: NCT05041647
Title: A Pilot, Double-Blind, Randomized, Placebo-Controlled Trial Evaluating the Efficacy and Safety of a Cannabis-Infused Oil For Treatment of Insomnia in Major Depression
Brief Title: Cannabinoids as a Treatment for Insomnia in Major Depression
Acronym: CANMDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Benicio Frey, Professor of Psychiatry and Behavioural Neurosciences, Prinicipal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CANMDD001
Record Dates: First submitted 2021-07-14; First posted 2021-09-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Depressive Disorder, Major; Sleep Disorder; Depression; Insomnia Chronic
Keywords: Mental Health; Cognition; Sleep Disorders; Major Depressive Disorder; Chronic Insomnia; Cannabis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major; Sleep Wake Disorders; Depression; Psychological Well-Being; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: The study will be a pilot, three-arm, randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants will be randomly assigned in a 1:1:1 manner to one of the three treatment arms using a computer-generated, permuted-block randomization schedule. Randomization will be stratified by sex. All of the treating physicians who will be also administering the clinical questionnaires, the trained research assistants conducting cognitive testing, as well as any other trial staff, will be blinded to the subjects' status until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High CBD [25:1] (Experimental): * 1 dose (1 mL) of HIGH CBD
  * 50 mg/ml CBD and 2 mg/ ml THC
  Interventions: Drug: 25:1 CBD/THC
- Low CBD [5:1] (Experimental): * 1 dose (1 mL) of LOW CBD
  * 10 mg/ml CBD and 2 mg/ ml THC
  Interventions: Drug: 5:1 CBD/THC
- Placebo (Placebo Comparator): * 1 dose (1 mL) of PLACEBO
  * No active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 25:1 CBD/THC — * 1 dose (1 mL) of HIGH CBD
  * 50 mg/ml CBD and 2 mg/ ml THC
  Other Names: High CBD
  Arms: High CBD [25:1]
Drug: 5:1 CBD/THC — * 1 dose (1 mL) of LOW CBD
  * 10 mg/ml CBD and 2 mg/ ml THC
  Other Names: Low CBD
  Arms: Low CBD [5:1]
Other: Placebo — * 1 dose (1 mL) of PLACEBO
  * No active ingredients
  Arms: Placebo

SUMMARY:
This single-site study is a pilot, three-armed, double-blinded, placebo-controlled randomized controlled trial (RCT) that will determine the feasibility of a definitive RCT investigating the use of cannabis oil as a treatment for insomnia in individuals with MDD. The study will also determine whether standard THC with higher CBD vs lower CBD has a differential impact on insomnia. The study will also analyze other important objective parameters of sleep including total sleep time and sleep efficiency from actigraphy data. Optional polysomnography data may also be collected and analyzed. In addition, standardized, validated instruments will be used to collect data on severity of depressive symptoms, cognitive functioning biological rhythm disruption, daytime sleepiness, health-related quality of life (HRQoL), healthcare resource utilization, work productivity and activity impairment, as well as other side effects, in order to better understand the potential impact of the use of cannabis oil on these important health outcomes.

DETAILED DESCRIPTION:
The study will be a three-arm, randomized, double-blind, placebo-controlled trial. The study population will include 60 males and females, ages 19 and older, who report chronic problems with insomnia at least three times per week for at least three months and have a diagnosis of co-morbid MDD. Eligible participants will complete a urine screen for drugs of abuse including opioids, cannabis, benzodiazepines and amphetamines before treatment randomization. Participants with a positive screen for any of these drugs of abuse will be excluded from the study. If the drug screen is negative, the principal investigator will assess patient health history and perform a physical examination. All study participants must be able to fully understand the study procedures and must sign a research ethics board (REB)-approved informed consent before study entry. A neuropsychological battery will be used to assess cognitive function in the domains of attention, verbal memory, psychomotor functioning, and executive functioning at baseline and at the end of the 4-week treatment in order to examine possible cognitive benefits or side effects from the treatment. These cognitive domains were chosen because these domains are known to be negatively affected by chronic insomnia and by cannabis use. Patients will also complete a series of clinician-rated and self-reported questionnaires.

During the 4-week treatment period, participants will be instructed to start treatment with a single, dose of oil at bedtime. Each dose will have either 50 mg/ml CBD and 2 mg/ml THC (High CBD arm; MLP-001) or 10 mg/ml CBD and 2 mg/ml THC (Low CBD arm; MLP-002). Non-responding study participants will add 1 additional dose to their respective treatment after 2 weeks if a higher dosage is needed based on an Insomnia Severity Index (ISI) reduction of >8 points and tolerability (side effects). Responding participants will continue with 1 dose of their treatment after 2 weeks. This dose range is based on previous studies showing that the effective dosage of THC to improve sleep ranged, on average, between 5 and 15 mg daily.

ELIGIBILITY:
Inclusion Criteria

1. Age 19 or above (A minimal age of 19 was chosen in order to align with the cannabis legalization rules of the Province of Ontario, where the research participants will be recruited from: https://www.ontario.ca/page/cannabis-legalization#section-1)
2. Diagnosis of MDD according to the Structured Clinical Interview for DSM-5 (SCID-5)
3. Diagnosis of Insomnia Disorder according to the Duke Structured Interview for Sleep Disorders Patient Health Questionnaire (PHQ-9) score of <10, indicating severity of mild-to-no depression (This criterion is important because a proper diagnosis of current co-morbid insomnia disorder cannot be accurately ascertained during acute major depressive episodes)
4. Participant must be willing and able to complete self-reported assessments, including having sufficient fluency in English
5. Participant must be willing to wear a wrist-worn actiwatch device
6. Participants may be using psychotropic medications for treatment of depression, except benzodiazepines or any other sleep aids, as long as the dosage remains the same from a minimum of 2 months prior to study enrolment until the end of the study (This criterion is important because many individuals with MDD use antidepressant agents and this criterion would make the results more generalizable and useful in real life clinical practice)

Exclusion Criteria

1. Lifetime diagnosis of Schizophrenia, Bipolar Disorder or any other psychotic disorder, as well as current or recent (last 6 months) Alcohol or Substance Use Disorder according to the SCID-5
2. Individuals with current diagnosis of Generalized Anxiety Disorder, Panic Disorder, Obsessive-Compulsive Disorder, Post-Traumatic Stress Disorder or Eating Disorder will be excluded because these psychiatric disorders are associated with sleep disturbance; however, because of the high rates of co-morbid psychiatric conditions in MDD lifetime/past diagnosis will be allowed in order for the results to be generalizable and useful in real life clinical practice
3. Current use of benzodiazepines or any other sleep aids
4. Positive screening for drugs of abuse including but not limited to opioids, cannabis, benzodiazepines, cocaine, and/or amphetamines (except prescribed stimulants for comorbid ADHD)
5. Presence of any sleep disorder other than insomnia that is considered the primary diagnosis, determined by the Duke Structured Interview for Sleep Disorders (e.g. Sleep Apnea, Limb Movement Disorder, or Circadian Rhythm Disorders)
6. Presence of unstable medical conditions
7. Pregnancy or breastfeeding (female participants will need to agree to use an acceptable contraceptive method during the study because of potential unknown teratogenic effects of cannabinoids
8. Allergy to cannabis or any components of the cannabis treatment (including terpenes)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 1 year, at the completion of the study
  Rates > 80% using descriptive statistics
Retention Rate | 1 year, at the completion of the study
  Rates > 80% using descriptive statistics

SECONDARY OUTCOMES:
Sleep onset latency and wake after sleep onset | through study completion, an average of 4 weeks
  Change in time (minutes) as measured using actigraphy
Treatment compliance | through study completion, an average of 4 weeks
  Completion rate > 80% using descriptive statistics

OTHER OUTCOMES:
Self-Reported Sleep Quality | through study completion, an average of 4 weeks
  A measure of self-reported sleep quality via questionnaires and sleep diaries
Cognitive Functioning | through study completion, an average of 4 weeks
  Battery of cognitive function that cover cognitive domains associated with insomnia and cannabis use.
Mean THC/CBD Dosing | through study completion, an average of 4 weeks
  Average THC and CBD dosage with the most optimal trade-off between efficacy and tolerability
Health-Related Quality of Life (HRQoL) | through study completion, an average of 4 weeks
  Short questionnaire to evaluate five dimensions of Health-Related Quality of Life
Healthcare Resource Utilization and Work Productivity | through study completion, an average of 4 weeks
  Short questionnaires to capture economic resource utilization and work productivity

CONTACTS AND LOCATIONS:
Overall Officials: Benicio N Frey, MD, MSc, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton; Nirushi Kuhathasan, PhD, Study Chair — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broyd SJ, van Hell HH, Beale C, Yucel M, Solowij N. Acute and Chronic Effects of Cannabinoids on Human Cognition-A Systematic Review. Biol Psychiatry. 2016 Apr 1;79(7):557-67. doi: 10.1016/j.biopsych.2015.12.002. Epub 2015 Dec 8. PMID 26858214
- [Background] Babson KA, Sottile J, Morabito D. Cannabis, Cannabinoids, and Sleep: a Review of the Literature. Curr Psychiatry Rep. 2017 Apr;19(4):23. doi: 10.1007/s11920-017-0775-9. PMID 28349316
- [Background] Gates PJ, Albertella L, Copeland J. The effects of cannabinoid administration on sleep: a systematic review of human studies. Sleep Med Rev. 2014 Dec;18(6):477-87. doi: 10.1016/j.smrv.2014.02.005. Epub 2014 Mar 7. PMID 24726015
- [Background] Kuhathasan N, Dufort A, MacKillop J, Gottschalk R, Minuzzi L, Frey BN. The use of cannabinoids for sleep: A critical review on clinical trials. Exp Clin Psychopharmacol. 2019 Aug;27(4):383-401. doi: 10.1037/pha0000285. Epub 2019 May 23. PMID 31120284